CLINICAL TRIAL: NCT06859320
Title: Outcomes Of Laparoscopic Sleeve Gastrectomy In Patients With Hypothyroidism And Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, faculty of medicine, Zagazig University, Egypt., Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #1108\25-Feb-2025
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity; hypothyroidism; Depression
MeSH Terms: conditions — Obesity; Hypothyroidism; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- morbid obesity and overweight in patients with hypothyroidism and depression (Other)
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — laparoscopic sleeve gastrectomy is one of the popular bariatric surgeries known for weight reduction

SUMMARY:
Sleeve gastrectomy (SG) continues to be one of the most popular bariatric procedures all over the world. It has been established that obesity is a predisposing factor for several comorbidities, including life-threatening conditions. Many studies have discussed the impact of sleeve gastrectomy on TSH level. But, since most obese patients have some sort of depression, we will try to study the impact of sleeve gastrectomy, depression and hypothyroidism on each other.

ELIGIBILITY:
Inclusion Criteria:

* obese patients with depression and hypothyroidism controlled by medical treatment candidate for sleeve gastrectomy

Exclusion Criteria:

* patients less than 18 or above 60
* other psychiatric or medical disorders.
* patients not fit for surgery
* un controlled patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
thyroid function tests | from one day to one year after surgery
  TSH,T3,T4 are measured pre and post operative
depression | from one day to one year after surgery
  depression status is compared pre-operative and post-operative using depression questionnaire (PHQ-9)( patient health questionnaire-9)
weight | from one day to one year after surgery
  weight of the patient will be measured in Kg using weight scale
dose of thyroid replacement therapy | monthly from one day to one year post surgery.
  the dose of L-thyroxin is monitored in microgrames
gasteric leakage | from one day to 1 week post-surgery
  leakage after surgery from staple line measured in ml in the drain
wound infection | from one day to 2 weeks post-surgery
  wound infection will be identified by pus in the drain or in the wound

SECONDARY OUTCOMES:
age | 2 days pre-operative
  age will be measured in years
sex | 2 days pre-operative
  sex of patient (male or female) will be recorded before surgery
BMI ( Body Mass Index) | 2 days before surgery to one year after surgery
  BMI is measured by the sum of weight in kg divided by the squared height in meters

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Zagazig, Sharqia Province
  - Zagazig University Hospitals, Zagazig